CLINICAL TRIAL: NCT01666912
Title: Etonogestrel-releasing Subdermal Implant for Adolescents in the Postpartum Period: a Randomized Controlled Trial
Brief Title: Postpartum Etonogestrel Implant for Adolescents
Acronym: PPImplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Amy Bryant, Assistant Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PPI-12-0732
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-03

CONDITIONS: Adolescence; Contraception; Postpartum
Keywords: adolescence; contraception; postpartum; rapid repeat pregnancy
MeSH Terms: interventions — Contraceptive Agents; etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6 week postpartum contraceptive implant (Active Comparator): randomized to receive contraceptive implant at normal 6 week postpartum visit
  Interventions: Drug: Contraceptive implant
- Immediate postpartum contraceptive implant (Experimental): randomized to receive contraceptive implant prior to leaving the hospital postpartum
  Interventions: Drug: Contraceptive implant

INTERVENTIONS:
Drug: Contraceptive implant
  Other Names: Implanon, Nexplanon, etonogestrel contraceptive implant

SUMMARY:
This is a prospective study comparing two groups of 48 adolescent women each. The intervention group will receive a contraceptive implant postpartum, prior to discharge from the hospital. The control group will receive a contraceptive implant at the usual 6 week postpartum clinic visit. During prenatal care, participants will be consented and screened for enrollment. After delivery, these women will be assessed and consented for enrollment into the study. Women who consent for enrollment will be randomized. Women will be followed up at 3 months, 6 months, 9 months, and 1 year after contraceptive implant insertion. At each follow up, women will be assessed for continuation of and satisfaction with this method of contraception.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents ages 14-24 attending prenatal care
* Greater than 20 weeks estimated gestational age
* English or Spanish-speaking
* Desire to use the contraceptive implant for contraception postpartum
* Anticipated delivery of a healthy infant vaginally or by cesarean.

Exclusion Criteria:

Participants will not be eligible for participation if they have any contraindications to contraceptive implant use, including

* current or past history of thrombosis or thromboembolic disorders
* hepatic tumors (benign or malignant)
* active liver disease
* undiagnosed abnormal genital bleeding
* known or suspected carcinoma of the breast (or a personal history of breast cancer)
* hypersensitivity to any of the components of the contraceptive implant.
* Current use of any medications known to induce hepatic enzymes, including but not limited to: barbiturates, bosentan, carbamazepine, felbamate, griseofulvin, oxcarbazepine, phenytoin, rifampin, St. John's wort, or topiramate

Characteristics that would preclude involvement after delivery:

* Birth of a stillborn infant.
* Maternal ICU admission after delivery
* Maternal postpartum hemorrhage requiring blood transfusion
* Prolonged hospital stay (>7 days) postpartum
* Coagulopathy associated with the pregnancy
* Severe pregnancy-induced hypertension
* Fever >38 degrees C postpartum
* Adolescent women who are not competent to consent, secondary to stress from the labor process, for example severe pain or sleep deprivation, will not be offered enrolment into the trial

Ages: 14 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2012-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina Hospitals, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 6 Week Postpartum Contraceptive Implant: randomized to receive contraceptive implant at normal 6 week postpartum visit
  Contraceptive implant
- Immediate Postpartum Contraceptive Implant: randomized to receive contraceptive implant prior to leaving the hospital postpartum
  Contraceptive implant
Period: Overall Study
Arm/Group | 6 Week Postpartum Contraceptive Implant | Immediate Postpartum Contraceptive Implant
Started | 48 | 48
Completed | 27 | 37
Not Completed | 21 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 Week Postpartum Contraceptive Implant | Immediate Postpartum Contraceptive Implant | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (2.58) | 21 (2.35) | 21 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 48 | 96
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 19 | 38
  Not Hispanic or Latino | 29 | 29 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 14 | 26
  White | 34 | 33 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 48 | 48 | 96

OUTCOME MEASURES:

1. Primary Outcome: Continuation at 1 Year
Description: The number of participants using the contraceptive implant at one year postpartum among women who have the implant placed immediately postpartum vs. at 6 weeks postpartum.
Time Frame: 12-14 months
Measure: Number; unit: participants
Arm/Group | 6 Week Postpartum Contraceptive Implant | Immediate Postpartum Contraceptive Implant
Number analyzed (Participants) | 27 | 37
participants | 21 | 30

2. Secondary Outcome: Satisfaction
Description: To assess satisfaction with the contraceptive implant inserted in the postpartum period, using a scale of 0-10, with 0 being "not satisfied at all" to 10 being "extremely satisfied."
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 6 Week Postpartum Contraceptive Implant | Immediate Postpartum Contraceptive Implant
Number analyzed (Participants) | 27 | 37
units on a scale | 8.68 (1.36) | 8.29 (2.14)

3. Secondary Outcome: Rapid Repeat Pregnancy
Description: To assess rapid repeat pregnancies among the study population, ie, the number of participants who reported a repeat pregnancy within 12 months postpartum.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | 6 Week Postpartum Contraceptive Implant | Immediate Postpartum Contraceptive Implant
Number analyzed (Participants) | 27 | 37
participants | 2 [1 to 5] | 5 [4 to 6]

ADVERSE EVENTS:
Arm/Group | 6 Week Postpartum Contraceptive Implant | Immediate Postpartum Contraceptive Implant
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes